CLINICAL TRIAL: NCT05852314
Title: Culturally Adapted Manual-Assisted Problem-Solving Intervention for Women With Suicidal Ideation in Postnatal Period in Pakistan: A Feasibility Trial
Brief Title: A Problem-Solving Intervention for Women With Suicidal Ideation During Postnatal Period in Pakistan
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CMAP- PNSI
Record Dates: First submitted 2023-05-01; First posted 2023-05-10 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Postnatal Depression
Keywords: Postnatal Depression; Suicidal Ideation; LMICs; CMAP
MeSH Terms: conditions — Depression, Postpartum; Suicidal Ideation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Culturally Adapted Manual Assisted Therapy (CMAP-SI) (Experimental): Participants in this arm will be offered the CMAP-SI intervention. The intervention will be delivered by trained researchers.
  Interventions: Behavioral: Culturally Adapted Manual Assisted Therapy (CMAP-SI)
- Treatment as Usual (TAU) (No Intervention): Local medical, psychiatric, and primary care services provide standard routine care in Pakistan. Participants will receive an initial assessment along with TAU as ascertained by their treating primary care physician (General Practitioner, GP). As part of the safety protocol, we will obtain the contact details of the participants GP. We will also obtain the details of any treatment received by each participant. Research psychologists delivering the interventions will not be involved with the participants allocated to the TAU.

INTERVENTIONS:
Behavioral: Culturally Adapted Manual Assisted Therapy (CMAP-SI) — C-MAP has been adapted from a self-help guide called Life After Self-Harm based on the principles of CBT. It is a brief problem-solving therapy comprising have 4 sessions weekly and then 4 fortnightly and last about 50 minutes each. The manual has been translated to Urdu giving special consideration to cultural adaptation of phrases and concepts to reflect Pakistani culture. Additionally, culturally appropriate case scenarios were incorporated and a consensual view to addressing cultural factors such as gender role, family conflicts and financial difficulties was taken. The culturally adapted intervention consists of the following components: evaluation of self-harm attempt, crisis skills, problem-solving and CBT techniques to manage emotions, negative thinking, interpersonal relationships, and relapse prevention strategies. Participants will receive sessions according to adapted CMAP-SI manual.
  Arms: Culturally Adapted Manual Assisted Therapy (CMAP-SI)

SUMMARY:
The aim of this study is to determine the feasibility and acceptability of culturally adapted CMAP for suicidal Ideation for women in postnatal period.

Objectives

1. To adapt existing CMAP Intervention for suicidal ideation (CMAP-SI) in postnatal period.
2. To investigate whether CMAP-SI is feasible and acceptable among women presenting suicidal Ideations in postnatal period; and
3. To test whether there is an indication for the effects of the CMAP in reducing suicidal thoughts among women in postnatal period.
4. To explore participants experiences with CMAP-SI Intervention.

DETAILED DESCRIPTION:
Suicide is a major public health concern globally, affecting not only the individuals but also family members and society through increased resource costs and productivity loss. Although suicides and suicide attempts occur at a lower rate during pregnancy and the postpartum period than in general population, the prevalence of suicidal thoughts during these periods ranges from 5-14% worldwide and this may result in suicide attempts and completions. There is a growing evidence suggesting that suicidal thoughts and behaviour among women in postnatal period in Low-and Middle-Income Countries (LMICs) are comparable to postnatal women in high resource settings. For instance, in observational studies based on hospital samples of women in postnatal period, 11% women had suicidal behaviour (i.e., thoughts and attempts) in Pakistan, 14% in Ethiopia and 13.6% in Nepal. The causes of these high prevalence rates point to the underlying maternal health issues such as antenatal depression and common mental disorders such as anxiety and depression. Evidence based interventions exists in prevention, care and treatment of suicidal thoughts such as Cognitive Behavioural Therapy (CBT). To deliver a CBT based intervention in Pakistani context, Husain and colleagues tailored a treatment manual: "Life after Self-Harm" to the general population in Pakistan. This Culturally Adapted Manual Assisted Problem solving (CMAP) aims at suicide prevention by reducing the probability of self-harm. Pakistan being a low resource setting faces a huge challenge to provide health care to its population. Therefore, it is important to screen women in postnatal period for risk for suicidal thoughts and behaviour, as well as, the maternal health problems. It is equally important to deliver culturally sensitive interventions which are addressing the psycho-social context wherein suicidal behaviour occurs. Thus, the main aim of this study is to determine the feasibility and acceptability of culturally adapted CMAP for suicidal Ideation for women in postnatal period.

ELIGIBILITY:
Inclusion Criteria:

1. 16 to 44-year-old mothers with children 0 - 30 months old
2. Residents of the trial site catchments area
3. Able to provide informed consent
4. Presenting with suicidal ideation as measured by the Beck Suicidal Ideation Scale (BSSI) (must score 1 or 2 on item 4 and 5)
5. Not requiring in-patient psychiatric treatment.

Exclusion Criteria:

We will exclude mothers with any physical or psychiatric condition severe enough to prevent study participation.

Ages: 16 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility and Acceptability | At 3 months after baseline
  The feasibility is defined as engagement with the intervention, its usability in daily life, as well as its potential for delivering a full trial in future. The feasibility of the study procedures will be assessed through monitoring recruitment and retention rates. Acceptability operationalised as the extent to which the participants receiving the intervention considered it to be appropriate, will be assessed through each participant's attendance rates in the intervention session. Additionally, the feasibility and acceptability will also be measured through qualitative interviews at post intervention

SECONDARY OUTCOMES:
Beck Scale for Suicidal Ideation (BSS) (Beck et al., 1988) | Baseline and 3 months
  Beck Scale for Suicidal Ideation will be used to measure the reduction in frequency and intensity of suicidal thoughts at baseline and at 3 months. The BSS is a 21-item measure assessing the severity of the suicidal ideation (Beck et al., 1988). Each item is scored from 0 to 2. The total score is obtained by adding the first 19 items and ranges from 0 to 38. High score represents high suicidal ideation. The BSS has good psychometric properties in English (Beck et al., 1988) This scale has been previously used in Pakistan (Husain et al., 2014) and the reported Cronbach's alpha for the Urdu translation of the BSI were 0.75 and 0.89 (Husain et al., 2014) respectively.
Suicide Attempt and Self-Harm (SASH) (Eylem, 2011) | Baseline and 3 months
  Suicide Attempt and Self-Harm consists of four questions measuring the previous suicide attempt and the presence of self-harm during last 6 weeks with a response on either 'yes, with a frequency of suicide attempt or self harm' or 'no'. SASH questions were taken from the original Self-Harm Questionnaire (Eylem, 2010). The original scale showed good psychometric properties (Eylem, 2010; Ougrin & Boege, 2013).
Edinburgh postnatal depression scale (EPDS) (Cox et al., 1987) | Baseline and 3 months
  Edinburgh postnatal depression scale will be used to screen depression in mothers with children aged 0-30 months. The maximum score of EPDS is 30, while score 10 or above shows possible depression. The EPDS has been translated into Urdu and validated in Pakistan (Husain et al., 2013).
Beck Depression Inventory (BDI) (Beck et al., 1961) | Baseline and 3 months
  Beck Depression Inventory will be used to measure symptoms of depression. BDI comprised of 21 items. Each item is scored from 0 to 3. The severity ranges from minimal depressed (score lower than 13) to severely depressed (scores between 29 and 63). It is a reliable and valid measure for assessing depression. The Cronbach's alpha for the Urdu translation of the instrument was 0.96 (Husain et al., 2014).
Life Events Checklist (Husain et al., 2000) | Baseline and 3 months
  Life events and difficulties will be assessed using a specially designed questionnaire based on our previous work in Pakistan. The domains that accounted for most of the life events and difficulties were included and rated categorically as present or not in the previous 12 months. This questionnaire has been used in a study of postnatal depression in rural Pakistan (Rahman, Iqbal, & Harrington, 2003) and for perinatal depression in Urban Pakistan (Husain et al., 2011).
Oslo- 3 Social Support Scale (O3SSS) (Dalgard, 2009) | Baseline and 3 months
  Oslo- 3 Social Support Scale will be used to assess the relationship with friends, family and neighbours. Each item is scored on a 5-point rating scale, and the total score ranges from 3 to 15, with high scores indicating a greater level of support. Its structure and reliability have not been well-documented despite its widespread use. The instrument has been validated in Urdu (Husain et al., 2012) and the Cronbach's alpha for the Urdu translation of the instrument was 0.46 (Husain et al., 2021).
Euro Quol (EQ-5D) (Rabin & Charro, 2001) | Baseline and 3 months
  Euro Quol -5D will be used to measure the health-related quality of life. EQ-5D is an instrument measuring health quality of life and has 5 items: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression (Rabin & Charro, 2001). Each item is required to be rated as 1 (no problem), 2 (some problem) or 3 (extreme problem). The current health state is also rated on a scale ranging from 0 (worst imaginable state) to 100 (best imaginable state). The instrument has been validated in Urdu (Husain et al., 2017).

CONTACTS AND LOCATIONS:
Overall Officials: Nasim Chaudhry, MD, Principal Investigator — Pakistan Institute of Living and Learning
Locations (1):
- Benazir Bhutto Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No